CLINICAL TRIAL: NCT07243483
Title: Prospective, Multicenter, Clinical-biological Cohort Study to Assess Pharmacokinetics and Pharmacodynamics (PK-PD) of Venetoclax (VEN) in Patients With Acute Myeloid Leukemia (AML)
Brief Title: Study of the Relationship Between the Pharmacokinetics (PK) and Pharmacodynamics of Venetoclax in Patients With Acute Myeloblastic Leukemia
Acronym: EUREKA-VEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Fédération Leucémie Espoir (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ET24-223
Record Dates: First submitted 2025-10-02; First posted 2025-11-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Pharmacokinetics; Venetoclax; Pharmacodynamics; Cytologic response; Azole antifungal
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Clinical-biological cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with acute myeloid leukaemia receiving venetoclax-azicitine as first line (Experimental): Blood samples
  Interventions: Other: Pharmacokinetic dosages of venetoclax

INTERVENTIONS:
Other: Pharmacokinetic dosages of venetoclax — Blood samples for pharmacokinetic dosing of venetoclax at different endpoints of treatment period

SUMMARY:
This is a prospective, multicenter, clinical-biological cohort study. Its objective is to assess the pharmacokinetics-pharmacodynamics (PK-PD) of venetoclax (VEN) in patients with Acute Myeloid Leukemia (AML).

This study involves only minimal risks and constraints related to the collection of biological samples (blood samples for PK testing) and the collection of clinical data. Therapeutic management of patients participating in this study is not changed. A total of 100 patients will be included in the study over a 12-month period. A maximum of 21 additional samples are planned, with a maximum of 12 mL of blood per sampling day (4 mL at each sampling time) for PK dosing of venetoclax.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged of at least 18 years on day of signing informed consent
* Patient with histologically-confirmed diagnosis of Acute Myeloblactic Leukaemia according to classification ELN 2022 (European Leukemia Net 2022)
* Patient who has to initiate treatment venetoclax-azacitidine as first line. Note : triple associations with targeted therapy are not authorized
* Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed.
* Patient must be affiliated or benificiary of a social security system.

Exclusion Criteria:

* Patient with acute promyelocytic leukemia (APL, AML3)
* Patient with AML eligible to intensive chemotherapy
* Patient previously treaed with venetoclax and/or azacitidine
* Patient participating to another clinical trial with a medicinal product
* Any condition that contraindicates blood sampling procedures required by the protocol
* Any psychological, family, geographical, or social situation that, according to investigator's judgment, could potentially prevent the signing of an informed consent form and/or woulld likely interfere compliance with study procedures.
* Patient under curatorship, guardianship or judicial protection
* Pregnant or breast-feeding female patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Best pharmacokinetic (PK) indicator of response to treatment in patients with AML - Biological endpoint | From the first day of venetoclax administration to end of the treatment (days)
  To assess PK exposure parameters : AUC (area under the curve) of venetoclax at steady state
Best pharmacokinetic (PK) indicator of response to treatment in patients with AML - Biological endpoint | From the first day of venetoclax administration to end of the treatment (days)
  To assess PK exposure parameters : Minimal Concentration (Cmin) of venetoclax at steady state
Best pharmacokinetic (PK) indicator of response to treatment in patients with AML - Biological endpoint | From the first day of venetoclax administration to end of the treatment (days)
  To assess PK exposure parameters : Peak Plasma Concentration (Cmax) of venetoclax at steady state
Best pharmacokinetic (PK) indicator of response to treatment in patients with AML - Biological endpoint | From the first day of venetoclax administration to end of the treatment (days)
  To assess PK exposure parameters : Equilibrium concentration (Css) of venetoclax at steady state
Best pharmacokinetic (PK) indicator of response to treatment in patients with AML - Clinical Endpoint | From the first day of venetoclax administration up to day 28 (end of the first venetoclax cure)
  Proportion of patients with a complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) or partial remission (PR) or no remission

SECONDARY OUTCOMES:
To assess relationship between different PK markers of venetoclax and its clinical efficacy. | From the first day of venetoclax administration and through study completion, at least 24 months
  Correlation between PK exposure parameters (including Cmin, Cmax, Css) of venetoclax and clinical outcome (cytologic response at cycle 6, survival without progression and overall survival).
To assess correlation between plasmatic exposition to venetoclax and occurrence of adverse events | From the the first day of venetoclax administration to the last day (Day 168) of venetoclax administration
  Correlation between PK exposure parameters (including Cmin, Cmax, Css) of venetoclax and occurence of adverse events grade equal or superior to 3 related to venetoclax/azacitidine and their impact on treatment administration
To assess inter-individual and intra-individual variability in plasma exposure to venetoclax. | From the first day of ventoclax administration and nd through study completion, at least 24 months
  Coefficient of variation of AUC and Cmin at steady state for venetoclax

OTHER OUTCOMES:
To assess the relationship between plasmatic venetoclax exposition and response to treatment | From the first day of venetoclax administration to through the study, at least 24 months
  To assess correlation between minimal concentration of venetoclax and minimal residual disease
To assess the relationship between plasmatic venetoclax exposition and response to treatment | From the first day of venetoclax administration to through the study, at least 24 months
  To assess correlation between Peak Plasma Concentration (Cmax) of venetoclax and minimal residual disease
To assess the relationship between plasmatic venetoclax exposition and response to treatment | From the first day of venetoclax administration to through the study, at least 24 months
  To assess correlation between Equilibrium concentration of venetoclax (Css) and minimal residual disease
To assess interaction between azole antifungals and venetoclax | From the the first day of venetoclax administration to the last day (Day 168) of venetoclax administration
  Number of patients treated or not treated by an azole antifungal

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Leon Berard, Lyon
  - CHU de Saint-Étienne, Saint-Etienne